CLINICAL TRIAL: NCT05890014
Title: Effects of Diet on Perinatal Mood and Cognition
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Daniel Lamport, Principle Investigator, Dr Daniel Lamport, University of Reading
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: UReading mothers study
Record Dates: First submitted 2023-05-25; First posted 2023-06-05 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Mood; Mothers; Healthy
Keywords: Cognition; Mood; Flavonoids; Diet; Postpartum; Blood pressure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The investigators who process, score and analyse data will be masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High flavonoid group (Experimental): Participants will be encouraged to consume 2 x flavonoid-rich food items per day from the following list of flavonoid-rich foods across 30-days, above what they already consume each day, typically.
  Orange juice (190 mls) Grapefruit juice (169mls) Dark chocolate (64g) Spinach (109g) Blueberry (64g) Strawberry (157g) Blackberry (81g) Blackcurrant (61g) Cherries (182g) Plums (90g) Black grapes (142g) Oranges (247g) Black olives (89g) Red grapes (339g)
  Interventions: Dietary Supplement: Flavonoid-rich diet
- Low flavonoid group (Experimental): Participants will be encouraged to consume 1 x flavonoid-rich food items per day from the following list of flavonoid-rich foods across 30-days, above what they already consume each day, typically.
  Orange juice (190 mls) Grapefruit juice (169mls) Dark chocolate (64g) Spinach (109g) Blueberry (64g) Strawberry (157g) Blackberry (81g) Blackcurrant (61g) Cherries (182g) Plums (90g) Black grapes (142g) Oranges (247g) Black olives (89g) Red grapes (339g)
  Interventions: Dietary Supplement: Flavonoid-rich diet
- Control (No Intervention): Participants will be given no instructions regarding adding food items to their diet. They will be encouraged to continue their diet as normal for 30-days.

INTERVENTIONS:
Dietary Supplement: Flavonoid-rich diet — Inclusion of foods rich in flavonoids.
  Arms: High flavonoid group; Low flavonoid group

SUMMARY:
The baby blues are a significant event which can occur immediately following childbirth and is a normal experience occurring in up to 76% of new mothers, characterised by mood swings, irritability and sadness typically lasting 10-14 days. Research suggests that the more severe and longer duration of the baby blues, the higher risk of later postnatal mood disorders. Therefore, this represents a critical period which could benefit from an intervention which may prevent symptom onset or an increase in the severity of mood disorders later in the postpartum.

Evidence suggests that consumption of flavonoid rich foods can improve physical health, mood and cognition. Prior research investigating flavonoid intervention in mothers in the first 6 months and 1 year postpartum found significant benefits to mood in the new mothers after daily flavonoid supplementation, showing promise for the management of mood in a key period for mothers, where risk of Postnatal Depression (PND) is high. The immediate postpartum also represents a period of cognitive changes reported to affect up to 80% of new mothers. In addition, women during this time are at an increased risk of high blood pressure and hypertension, which is thought to be a risk factor for the onset and severity of depressive symptoms and cognitive decrements. Flavonoids have been reported to improve cognition and cardiovascular health, therefore, introducing a flavonoid intervention could have benefits to cognition and blood pressure in new mothers.

The aim of the current study will be to explore whether the implementation of a high flavonoid diet across a 30-day period will positively affect maternal mental health, cognition and blood pressure. Participants will be assigned to one of three groups; high or low flavonoid diet or a control condition for 30-days, starting at days 0-4 after birth. They will have visits from the researcher at 6 separate time points between the third trimester and 12 weeks postpartum. At each visit, participants will be asked to complete mood questionnaires (PANAS-NOW), Edinburgh Postnatal Depression Scale (EPDS), Postpartum Specific Anxiety Scale (PSAS), State-Trait Anxiety Inventory (STAI), Edinburgh Postnatal Depression Scale- Partner (EPDS-P) followed by a cognitive battery (MANT, RAVLT, PRMQ) and blood pressure recordings (systolic and diastolic blood pressure). Between visits, participants will be contacted by the researcher to record retrospective 24hr food recalls (Intake24).

DETAILED DESCRIPTION:
The study will employ a between-groups, randomised, controlled, participant-blind design with three groups and six time points. Participants will be allocated to one of three groups; a high flavonoid condition (consumption of 2 portions of flavonoid rich food per day), low flavonoid condition (consumption of one portion of flavonoid rich food per day) and a control (no change to diet). Participants will be quasi-randomised to condition based on their baseline flavonoid intake, taken at Timepoint 1 using the European Prospective Investigation of Cancer (EPIC)-Norfolk Food Frequency Questionnaire to ensure there is an even spread of baseline flavonoid consumption in participants across all conditions. At this timepoint, participants will additionally complete the Immediate Mood Scaler. Participants will be recruited at any stage of their pregnancy though testing will not take place until their third trimester (weeks 27+). Participants will be invited to a study investigating diet mood and cognition. The study will take place in person, at participant homes over 6 time points; 1) a screening session, 2) time 1 (third trimester), 3) time 2 (after birth 0-4 days, pre intervention), 4) time 3 (mid-way through intervention ~15 days), 5) time 4 (post-intervention ~30 days) and 6) time 5 (follow up, 12 weeks postpartum).

Interested participants will be invited to an in-person screening session. Once participants have consented to taking part, they will be asked to provide some demographic information (e.g. age, occupation, health or psychological diagnosis). Participants will then complete practice versions of the cognitive tests. At each timepoint, the experimenter will visit participants to complete outcome measures (PANAS-NOW, EPDS, PSAS, STAI, EPDS-P, MANT, Spatial n-back, RAVLT and PRMQ, Systolic and Diastolic blood pressure). Over the course of the study, participants will be contacted at nine random timepoints to complete retrospective 24hr food recalls using the software Intake24.

Participants in the flavonoid intervention groups will be contacted by the researcher shortly before time 2 where they will be sent a list of the intervention foods and asked to choose a food item which the researcher will bring to the testing session. This is to ensure that participants can start the intervention after the testing session at time 2 without needing to visit a supermarket during this sensitive time. During this session, participants will also be asked some questions about the baby and birth experience (e.g. how old their infant is, infants sex, mode of delivery, birth complications). After the outcome measures have been taken, participants will be informed of their condition and instructed to begin the intervention. The two intervention groups will also be asked to keep a food log of their selected intervention foods for the 30-day period.

At the final timepoint, upon completion of outcome measures, participants will receive the debrief document and they will receive information about payment and dietary assessment via email. Participants will also be reminded of their right to withdraw their data from the study if they wish. Helplines and support web links will be provided to all participants as well as encouragement for participants to contact their General Practitioner should they wish to seek support. Helplines and weblinks include Samaritans United Kingdom and PANDAS Foundation. Weblinks to National Health Service (NHS), MIND mental health charity and the Association for Postnatal Illness.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be pregnant (reliant on mothers' self-reporting)

Exclusion Criteria:

* Participants beyond 38 weeks of their pregnancy (reliant on mothers' self reporting)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03-14 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Mean depressive symptoms | Days 0-4 postpartum
  Assessed using scores from the Edinburgh Postnatal Depression Scale measure. Higher scores indicate higher levels of depressive symptoms. This questionnaire contains 10 items where participants rate how they have been feeling over the past 7 days on a 4-point Likert scale. Scores on this scale fall between 0-30 where higher scores indicate worse outcomes. The EPDS was designed for women who are pregnant or have just had a baby and has shown to be an efficient and effective way of identifying patients at risk for perinatal depression. This measure is suitable for use in new mothers and fathers.
Mean depressive symptoms | 2 weeks postpartum
  Assessed using scores from the Edinburgh Postnatal Depression Scale measure. Higher scores indicate higher levels of depressive symptoms. This questionnaire contains 10 items where participants rate how they have been feeling over the past 7 days on a 4-point Likert scale. Scores on this scale fall between 0-30 where higher scores indicate worse outcomes. The EPDS was designed for women who are pregnant or have just had a baby and has shown to be an efficient and effective way of identifying patients at risk for perinatal depression. This measure is suitable for use in new mothers and fathers.
Mean depressive symptoms | 4 weeks postpartum
  Assessed using scores from the Edinburgh Postnatal Depression Scale measure. Higher scores indicate higher levels of depressive symptoms. This questionnaire contains 10 items where participants rate how they have been feeling over the past 7 days on a 4-point Likert scale. Scores on this scale fall between 0-30 where higher scores indicate worse outcomes. The EPDS was designed for women who are pregnant or have just had a baby and has shown to be an efficient and effective way of identifying patients at risk for perinatal depression. This measure is suitable for use in new mothers and fathers.
Mean depressive symptoms | 12 weeks postpartum
  Assessed using scores from the Edinburgh Postnatal Depression Scale measure. Higher scores indicate higher levels of depressive symptoms. This questionnaire contains 10 items where participants rate how they have been feeling over the past 7 days on a 4-point Likert scale. Scores on this scale fall between 0-30 where higher scores indicate worse outcomes. The EPDS was designed for women who are pregnant or have just had a baby and has shown to be an efficient and effective way of identifying patients at risk for perinatal depression. This measure is suitable for use in new mothers and fathers.
Mean state anxiety | Days 0-4 postpartum
  Assessed using scores from the State-Trait Anxiety Inventory- State scale. Higher scores indicate higher levels of anxiety. This questionnaire is a measure of state and trait anxiety containing 40 items in total (20 for trait; 20 for state). Only the state scale (20 items) will be used in current research to measure situational anxiety. Participants are asked to agree or disagree with anxiety-related statements on a scale of 1-4 where higher scores indicate worse outcomes.
Mean state anxiety | 2 weeks postpartum
  Assessed using scores from the State-Trait Anxiety Inventory- State scale. Higher scores indicate higher levels of anxiety. This questionnaire is a measure of state and trait anxiety containing 40 items in total (20 for trait; 20 for state). Only the state scale (20 items) will be used in current research to measure situational anxiety. Participants are asked to agree or disagree with anxiety-related statements on a scale of 1-4 where higher scores indicate worse outcomes.
Mean state anxiety | 4 weeks postpartum
  Assessed using scores from the State-Trait Anxiety Inventory- State scale. Higher scores indicate higher levels of anxiety. This questionnaire is a measure of state and trait anxiety containing 40 items in total (20 for trait; 20 for state). Only the state scale (20 items) will be used in current research to measure situational anxiety. Participants are asked to agree or disagree with anxiety-related statements on a scale of 1-4 where higher scores indicate worse outcomes.
Mean state anxiety | 12 weeks postpartum
  Assessed using scores from the State-Trait Anxiety Inventory- State scale. Higher scores indicate higher levels of anxiety. This questionnaire is a measure of state and trait anxiety containing 40 items in total (20 for trait; 20 for state). Only the state scale (20 items) will be used in current research to measure situational anxiety. Participants are asked to agree or disagree with anxiety-related statements on a scale of 1-4 where higher scores indicate worse outcomes.

SECONDARY OUTCOMES:
Mean postpartum-specific anxiety symptoms | Days 0-4 postpartum
  Assessed using scores from the Postpartum-Specific Anxiety Scale. This is a 51-item questionnaire that examines the frequency of maternal and infant focused anxieties experienced by women over the last week. It can be used at any time during the first year following birth and is found to be a valid and reliable measure. Each response is given a score of between 1 and 4 with the maximum score being a total of 204, with higher scores indicating higher levels of anxiety where a score of 112 or above indicating likelihood the individual suffering from an anxiety disorder.
Mean postpartum-specific anxiety symptoms | 2 weeks postpartum
  Assessed using scores from the Postpartum-Specific Anxiety Scale. This is a 51-item questionnaire that examines the frequency of maternal and infant focused anxieties experienced by women over the last week. It can be used at any time during the first year following birth and is found to be a valid and reliable measure. Each response is given a score of between 1 and 4 with the maximum score being a total of 204, with higher scores indicating higher levels of anxiety where a score of 112 or above indicating likelihood the individual suffering from an anxiety disorder.
Mean postpartum-specific anxiety symptoms | 4 weeks postpartum
  Assessed using scores from the Postpartum-Specific Anxiety Scale. This is a 51-item questionnaire that examines the frequency of maternal and infant focused anxieties experienced by women over the last week. It can be used at any time during the first year following birth and is found to be a valid and reliable measure. Each response is given a score of between 1 and 4 with the maximum score being a total of 204, with higher scores indicating higher levels of anxiety where a score of 112 or above indicating likelihood the individual suffering from an anxiety disorder.
Mean postpartum-specific anxiety symptoms | 12 weeks postpartum
  Assessed using scores from the Postpartum-Specific Anxiety Scale. This is a 51-item questionnaire that examines the frequency of maternal and infant focused anxieties experienced by women over the last week. It can be used at any time during the first year following birth and is found to be a valid and reliable measure. Each response is given a score of between 1 and 4 with the maximum score being a total of 204, with higher scores indicating higher levels of anxiety where a score of 112 or above indicating likelihood the individual suffering from an anxiety disorder.
Mean current affect | Days 0-4 postpartum
  Assessed using scores from the Positive and Negative Affect Scale. This questionnaire has 20 items that describe some feelings and emotions. The participant needs to mark how much they are experiencing these feelings on a scale from 1-5. This produces scores of Positive Affect and Negative Affect; higher scores reflect higher positive or negative mood, respectively.
Mean current affect | 2 weeks postpartum
  Assessed using scores from the Positive and Negative Affect Scale. This questionnaire has 20 items that describe some feelings and emotions. The participant needs to mark how much they are experiencing these feelings on a scale from 1-5. This produces scores of Positive Affect and Negative Affect; higher scores reflect higher positive or negative mood, respectively.
Mean current affect | 4 weeks postpartum
  Assessed using scores from the Positive and Negative Affect Scale. This questionnaire has 20 items that describe some feelings and emotions. The participant needs to mark how much they are experiencing these feelings on a scale from 1-5. This produces scores of Positive Affect and Negative Affect; higher scores reflect higher positive or negative mood, respectively.
Mean current affect | 12 weeks postpartum
  Assessed using scores from the Positive and Negative Affect Scale. This questionnaire has 20 items that describe some feelings and emotions. The participant needs to mark how much they are experiencing these feelings on a scale from 1-5. This produces scores of Positive Affect and Negative Affect; higher scores reflect higher positive or negative mood, respectively.
Mean partner depressive symptoms | 0-4 postpartum
  Using the EPDS-P. This is a 10-item measure adapted from the EPDS. The EPDS-P is a revision of the EPDS to provide a proxy of the partners symptoms of depression, in this study, the mothers will complete the EPDS-P to provide information about paternal depressive symptoms. The scale and scoring of the EPDS-P is the same as the EPDS, though there is no cut-off in the EPDS-P to indicate likelihood for depressive disorder.
Mean partner depressive symptoms | 2 weeks postpartum
  Using the EPDS-P. This is a 10-item measure adapted from the EPDS. The EPDS-P is a revision of the EPDS to provide a proxy of the partners symptoms of depression, in this study, the mothers will complete the EPDS-P to provide information about paternal depressive symptoms. The scale and scoring of the EPDS-P is the same as the EPDS, though there is no cut-off in the EPDS-P to indicate likelihood for depressive disorder.
Mean partner depressive symptoms | 4 weeks postpartum
  Using the EPDS-P. This is a 10-item measure adapted from the EPDS. The EPDS-P is a revision of the EPDS to provide a proxy of the partners symptoms of depression, in this study, the mothers will complete the EPDS-P to provide information about paternal depressive symptoms. The scale and scoring of the EPDS-P is the same as the EPDS, though there is no cut-off in the EPDS-P to indicate likelihood for depressive disorder.
Mean partner depressive symptoms | 12 weeks postpartum
  Using the EPDS-P. This is a 10-item measure adapted from the EPDS. The EPDS-P is a revision of the EPDS to provide a proxy of the partners symptoms of depression, in this study, the mothers will complete the EPDS-P to provide information about paternal depressive symptoms. The scale and scoring of the EPDS-P is the same as the EPDS, though there is no cut-off in the EPDS-P to indicate likelihood for depressive disorder.
Mean subjective memory scores | Days 0-4 postpartum
  Prospective and retrospective memory questionnaire. The PRMQ is a 16-item rating scale, designed to assess the frequency of different types of memory failures whereby higher scores indicate greater frequency of memory failures. Participants are asked to score questions of a 5-point scale 1 (never), 2 (rarely), 3 (sometimes), 4 (quite often), 5 (very often). Results can be derived for prospective or retrospective, short-term or long-term, self-cued or environmentally cued.
Mean subjective memory scores | 2 weeks postpartum
  Prospective and retrospective memory questionnaire. The PRMQ is a 16-item rating scale, designed to assess the frequency of different types of memory failures whereby higher scores indicate greater frequency of memory failures. Participants are asked to score questions of a 5-point scale 1 (never), 2 (rarely), 3 (sometimes), 4 (quite often), 5 (very often). Results can be derived for prospective or retrospective, short-term or long-term, self-cued or environmentally cued.
Mean subjective memory scores | 4 weeks postpartum
  Prospective and retrospective memory questionnaire. The PRMQ is a 16-item rating scale, designed to assess the frequency of different types of memory failures whereby higher scores indicate greater frequency of memory failures. Participants are asked to score questions of a 5-point scale 1 (never), 2 (rarely), 3 (sometimes), 4 (quite often), 5 (very often). Results can be derived for prospective or retrospective, short-term or long-term, self-cued or environmentally cued.
Mean subjective memory scores | 12 weeks postpartum
  Prospective and retrospective memory questionnaire. The PRMQ is a 16-item rating scale, designed to assess the frequency of different types of memory failures whereby higher scores indicate greater frequency of memory failures. Participants are asked to score questions of a 5-point scale 1 (never), 2 (rarely), 3 (sometimes), 4 (quite often), 5 (very often). Results can be derived for prospective or retrospective, short-term or long-term, self-cued or environmentally cued.
Mean subjective mood scores | Baseline only
  Immediate mood scale-This questionnaire contains 22 items developed to assess dynamic components of mood. Participants are asked to rate their current mood state on a continuum using 7-point Likert scales (e.g., happy-sad, distracted-focused, sleepy-alert). For each item, an integer score between 1 and 7 is derived. The total score for this scale is the sum of the scores on all 22 items.
Subjective sleep scores | Days 0-4 postpartum
  Using the Pittsburgh Sleep Quality Index (PSQI). The PSQI is a validated measure of sleep assessing qualities and patterns within the last month of sleep habits in adults. Seven components of sleep (quality, latency, duration, efficiency, disturbance, use of sleep medication, daytime dysfunction) will be summed to achieve a global PSQI score ranging from 0 to 21 points, where scores above 5 indicates sleep problems.
Subjective sleep scores | 2 weeks postpartum
  Using the Pittsburgh Sleep Quality Index (PSQI). The PSQI is a validated measure of sleep assessing qualities and patterns within the last month of sleep habits in adults. Seven components of sleep (quality, latency, duration, efficiency, disturbance, use of sleep medication, daytime dysfunction) will be summed to achieve a global PSQI score ranging from 0 to 21 points, where scores above 5 indicates sleep problems.
Subjective sleep scores | 4 weeks postpartum
  Using the Pittsburgh Sleep Quality Index (PSQI). The PSQI is a validated measure of sleep assessing qualities and patterns within the last month of sleep habits in adults. Seven components of sleep (quality, latency, duration, efficiency, disturbance, use of sleep medication, daytime dysfunction) will be summed to achieve a global PSQI score ranging from 0 to 21 points, where scores above 5 indicates sleep problems.
Subjective sleep scores | 12 weeks postpartum
  Using the Pittsburgh Sleep Quality Index (PSQI). The PSQI is a validated measure of sleep assessing qualities and patterns within the last month of sleep habits in adults. Seven components of sleep (quality, latency, duration, efficiency, disturbance, use of sleep medication, daytime dysfunction) will be summed to achieve a global PSQI score ranging from 0 to 21 points, where scores above 5 indicates sleep problems.
Blood pressure | Days 0-4 postpartum
  Resting systolic and diastolic blood pressure will be taken with an ambulatory blood pressure monitor. Measurements will be taken on participants left arm and the mean of three consecutive measurements will be calculated.
Blood pressure | 2 weeks postpartum
  Resting systolic and diastolic blood pressure will be taken with an ambulatory blood pressure monitor. Measurements will be taken on participants left arm and the mean of three consecutive measurements will be calculated.
Blood pressure | 4 weeks postpartum
  Resting systolic and diastolic blood pressure will be taken with an ambulatory blood pressure monitor. Measurements will be taken on participants left arm and the mean of three consecutive measurements will be calculated.
Blood pressure | 12 weeks postpartum
  Resting systolic and diastolic blood pressure will be taken with an ambulatory blood pressure monitor. Measurements will be taken on participants left arm and the mean of three consecutive measurements will be calculated.
Verbal memory | Days 0-4 postpartum
  Assessed using the Rey Auditory Verbal Learning Test.
Verbal memory | 2 weeks postpartum
  Assessed using the Rey Auditory Verbal Learning Test.
Verbal memory | 4 weeks postpartum
  Assessed using the Rey Auditory Verbal Learning Test.
Verbal memory | 12 weeks postpartum
  Assessed using the Rey Auditory Verbal Learning Test.
Sustained attention and executive functioning | Days 0-4 postpartum
  Assessed with the Modified Attention Network Task with accuracy and reaction time as outcome measures.
Sustained attention and executive functioning | 2 weeks postpartum
  Assessed with the Modified Attention Network Task with accuracy and reaction time as outcome measures.
Sustained attention and executive functioning | 4 weeks postpartum
  Assessed with the Modified Attention Network Task with accuracy and reaction time as outcome measures.
Sustained attention and executive functioning | 12 weeks postpartum
  Assessed with the Modified Attention Network Task with accuracy and reaction time as outcome measures.
Visuospatial working memory | Days 0-4 postpartum
  Measured using the Visuospatial n-back with accuracy and reaction time as outcome measures.
Visuospatial working memory | 2 weeks postpartum
  Measured using the Visuospatial n-back with accuracy and reaction time as outcome measures.
Visuospatial working memory | 4 weeks postpartum
  Measured using the Visuospatial n-back with accuracy and reaction time as outcome measures.
Visuospatial working memory | 12 weeks postpartum
  Measured using the Visuospatial n-back with accuracy and reaction time as outcome measures.

OTHER OUTCOMES:
General diet | Baseline only
  Participants will complete a food frequency questionnaire at baseline using the EPIC Food Frequency Questionnaire. This measures contains a list of foods/drinks and the participant needs to state how often they consume each food/drink to assess participants' general diet.
24-hr dietary recall | Pregnancy (up to 10 weeks before birth date)
  Measured using Intake24. This tool will contact participants asking to provide details of all the foods consumed in the previous 24-hours.The participants can do this from their phone via weblink whereby participants self-report the food they consumed, time eaten, food portion sizes and preparation in addition to any dietary supplements. This timeframe will include three measures of 24hr recall (2 weekday and 1 weekend recording).
24-hr dietary recall | Postpartum during intervention (up to 34 days after birth)
  Measured using Intake24. This tool will contact participants asking to provide details of all the foods consumed in the previous 24-hours.The participants can do this from their phone via weblink whereby participants self-report the food they consumed, time eaten, food portion sizes and preparation in addition to any dietary supplements. This timeframe will include three measures of 24hr recall (2 weekday and 1 weekend recording).
24-hr dietary recall | Postpartum after intervention (up to 12 weeks after birth)
  Measured using Intake24. This tool will contact participants asking to provide details of all the foods consumed in the previous 24-hours.The participants can do this from their phone via weblink whereby participants self-report the food they consumed, time eaten, food portion sizes and preparation in addition to any dietary supplements. This timeframe will include three measures of 24hr recall (2 weekday and 1 weekend recording).

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Lamport, PhD, Principal Investigator — University of Reading
Locations (1):
- University of Reading, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data may be made available on a platform such as Open Science Framework (www.osf.io) or a data repository linked to academic journals, in accordance with Open Science principles.